CLINICAL TRIAL: NCT06805968
Title: Acute Effects of High Intensity Aerobic Exercise on Respiratory Function and Cognitive Status in Smoker Healthcare Workers
Brief Title: Effect of Exercise on Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Istanbul Gedik University (Other)
Responsible Party: Principal Investigator, ebrar atak, Asst. Prof., Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E56365223-050.02.02.2023.13754
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2023-09

CONDITIONS: Smokers
Keywords: smoker; aerobic; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- high-intensity aerobic exercise group (Experimental)
  Interventions: Other: High Intensity Exercise + Placebo
- low-intensity aerobic exercise group (Active Comparator)
  Interventions: Other: Low Intensity Exercise + Placebo

INTERVENTIONS:
Other: High Intensity Exercise + Placebo — high intensity exercise
  Arms: high-intensity aerobic exercise group
Other: Low Intensity Exercise + Placebo — low intensity exercise
  Arms: low-intensity aerobic exercise group

SUMMARY:
When we look at the literature, although 202 results are found when "high intensity training" AND "aerobic" is written in the PUBMED database, 27 to 86 results are found when "high intensity training" AND "cognitive" and "high intensity training" AND "respiratory" are written and searched. 5 results are found when "high intensity training" AND "smoking" is searched, but there is no study investigating cognitive and respiratory functions, and no results are found when "high intensity training" AND "smoker" is searched. As far as is known, there is no study investigating the acute effect of high intensity aerobic exercise on respiratory functions and cognitive status in special education personnel who smoke. We aim to contribute to the literature with this original aspect of our study.

DETAILED DESCRIPTION:
Primary objective: The primary objective of the study is to investigate the acute effects of high-intensity aerobic exercise on respiratory functions in special education personnel who smoke.

Secondary objective: The secondary objective of the study is to investigate the acute effects of high-intensity aerobic exercise on cognitive status in special education personnel who smoke.

Study questions

* Is there an acute effect of high-intensity aerobic exercise on respiratory functions in special education personnel who smoke?
* Is there an acute effect of high-intensity aerobic exercise on cognitive status in special education personnel who smoke?

Study Hypotheses:

H0: There is no acute effect of high-intensity aerobic exercise on respiratory functions in special education personnel who smoke.

H1: There is an acute effect of high-intensity aerobic exercise on respiratory functions in special education personnel who smoke.

H2: There is no acute effect of high-intensity aerobic exercise on cognitive status in special education personnel who smoke.

H3: High-intensity aerobic exercise has an acute effect on cognitive status in special education personnel who smoke.

H4: High-intensity aerobic exercise has a greater acute effect on respiratory function and cognitive status in special education personnel who smoke than low-intensity training.

H5: High-intensity aerobic exercise has a less acute effect on respiratory function and cognitive status in special education personnel who smoke than low-intensity training.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Participating in the Fageström Nicotine Dependence Questionnaire
* No comorbidities
* No comorbid diseases related to the orthopedic, neurological, cardiopulmonary system
* Participants who have not participated in another clinical trial in the last month

Exclusion Criteria:

* Participants who have had orthopedic and cardiopulmonary surgery in the last year
* Those with cardiac or pulmonary system disease
* Having sensory loss
* Participants with leg length inequality

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-09-03 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Smoking dependence level measurement | Duration of change in 1 day.
  Meausered with Fagerström Nicotine Dependence Questionnaire (FNBA)
FVC Measurement | Duration of change in 1 day.
  Respiratory Function Test. The COSMED microQuark spirometer used. Lung volume was evaluated.
FEV1 Measurement | Duration of change in 1 day.
  Respiratory Function Test. The COSMED microQuark spirometer used. Lung volume was evaluated.

SECONDARY OUTCOMES:
Cognitive status measurement with MOCA | Duration of change in 1 day.
  Measured with Montreal Cognitive Function Assessment Scale (MOCA)
Cognitive status measurement with Stroop Test | Duration of change in 1 day.
  Measured with Stroop Test

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Gedik University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided